CLINICAL TRIAL: NCT04725136
Title: A Phase I/IIa Clinical Trial to Evaluate the Safety and Explore the Efficacy of Multiple Doses of FURESTEM-AD Inj. for Moderate to Severe Chronic Atopic Dermatitis
Brief Title: Safety and Explore the Efficacy of Multiple Doses of FURESTEM-AD Inj. for Moderate to Severe Chronic Atopic Dermatitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K0104
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Atopic Dermatitis
Keywords: hUCB-MSC; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- High-dose repeat administration group (Experimental): FURESTEM-AD Inj 1.0 x 10^8 cells /body 3 repeated subcutaneous injection at 4 week intervals
  Interventions: Biological: FURESTEM-AD inj
- High-dose single administration group (Experimental): FURESTEM-AD Inj 1.0 x 10^8 cells /body 1 single subcutaneous injection, and Placebo 2 repeated subcutaneous injection at 4 week intervals
  Interventions: Biological: FURESTEM-AD inj
- Low-dose repeat administration group (Experimental): FURESTEM-AD Inj 5.0 x 10^7 cells /body 3 repeated subcutaneous injection at 4 week intervals
  Interventions: Biological: FURESTEM-AD inj
- Low-dose single administration group (Experimental): FURESTEM-AD Inj 5.0 x 10^7 cells /body 1 single subcutaneous injection, and Placebo 2 repeated subcutaneous injection at 4 week intervals
  Interventions: Biological: FURESTEM-AD inj
- Placebo (Placebo Comparator): Normal saline(0.9% NaCl) 3 repeated subcutaneous injection at 4 week intervals
  Interventions: Biological: FURESTEM-AD inj

INTERVENTIONS:
Biological: FURESTEM-AD inj — Repeated administration group: 3 times high or low dose at 4 week intervals. Single administration group: 1 time high or low dose, 2 times placebo injection at 4 week intervals Placebo: 3 times placebo injection at 4 week intervals.

SUMMARY:
A Phase I/IIa Clinical Trial to Evaluate the Safety and Explore the Efficacy of Multiple Doses of FURESTEM-AD inj. for Moderate to Severe Chronic Atopic Dermatitis

DETAILED DESCRIPTION:
Phase 1: Multicenter, repeated administration, disclosure, dose escalation, Evaluate safety and tolerability and explore efficacy

Phase 2a: Multicenter, repeated administration, random assignment, double blinding, parallel, Efficacy and safety are evaluated for repeated administration compared to placebo and single administration.

ELIGIBILITY:
Inclusion Criteria:

1. Of either gender, aged >=19
2. Atopic Dermatitis subjects who are coincident with Hanifin and Rajka diagnosis criteria
3. Chronic Atopic Dermatitis that has been present for at least 3 years
4. EASI>=16 at screening and baseline visit
5. IGA>=3, SCORAD index>=25, BSA >=10% of AD involvement at screegning and baseline visit
6. Subjects with documented record of inadequate response to the stable use of topical atopic dermatitis treatment within 24 weeks before participating in the study, or whom are inadvisable due to safety risks
7. Subjects who understand and voluntarily sign an informed consent form

Exclusion Criteria:

1. Subjects with medical history or surgery/procedure history
2. Subjects with diseases at the time of participation in this study (systemic infection, other serious skin disorders, pigmentation or extensive scarring in atopic dermatitis symptom region)
3. Renal dysfunction with creatinine >2.0 mg/dL at screening
4. Hepatic dysfunction with ALT or AST levels 2.5 times higher than the normal range at screening
5. ALC<800/mm3 at screening
6. Subjects with live vaccine administration within 12 weeks before baseline
7. Receipt of leukotriene receptor antagonists, systemic steroids, systemic or topical antihistamines, phototherapy, or systemic immunosuppressants/modulators including janus kinase (JAK) inhibitors, and/or any other systemic therapy within 4 weeks before Baseline
8. Receipt of topical steroids(class1~6), topical tacrolimus or pimecrolimus within 2 weeks before Baseline
9. Subjects who need prohibited medication during clinical period
10. Pregnant, breast-feeding women or women who plan to become pregnant during this study
11. Subjects who currently participate in other clinical trial or participated in other clinical trial within 4 weeks
12. Subjects with experience of administering FURESTEM-AD inj.
13. Any other condition which the investigator judges would make patient unsuitable for study participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | 24 weeks follow-up after first treatment
  safety information including drug tolerability

SECONDARY OUTCOMES:
Percentage of subjects whose EASI decreased by 50% or more at each evaluation visit compared to the baseline (EASI-50) | 24 weeks follow-up after first treatment
Percentage of subjects whose Eczema Area and Severity Index (EASI) was decreased from baseline by more than 75% at each visit (EASI-75) | 24 weeks follow-up after first treatment
Rate of change and Change in EASI from baseline | 24 weeks follow-up after first treatment
  EASI range is from 0 (clear) to 72 (severe)
Percentage of subjects whose Investigator's Global Assessment (IGA) score at each visit is 0 or 1 | 24 weeks follow-up after first treatment
  IGA score is from 0 (clear) to 5 (severe)
Percentage of subjects whose IGA at each visit is 0 or 1, or improved to 2 or higher | 24 weeks follow-up after first treatment
  IGA score is from 0 (clear) to 5 (severe)
Percentage of subjects whose SCORing Atopic Dermatitis (SCORAD) INDEX was decreased from baseline by more than 50% at each visit (SCORAD-50) | 24 weeks follow-up after first treatment
Rate of change and Change in SCORAD index from baseline at each visit | 24 weeks follow-up after first treatment
  SCORAD index range is from 0 (clear) to 103 (severe)
Change and rate of change in Body Surface Area (BSA) | 24 weeks follow-up after first treatment
Change and rate of change in total serum Immunoglobulin E (IgE) | 24 weeks follow-up after first treatment
Change and rate of change in Cytokine | 24 weeks follow-up after first treatment
  CCL17(TARC), CCL18(PARC), CCL26(eotaxin-3), CCL27(CTACK), IL-4, IL-17A, IL-22, SCCA2
Change and rate of change DLQI | 24 weeks follow-up after first treatment
Change and rate of change POEM | 24 weeks follow-up after first treatment
Change and rate of change Peak Pruritus NRS | 24 weeks follow-up after first treatment
Change and rate of change eosinophil | 24 weeks follow-up after first treatment
Use the number and total amount of rescue | 24 weeks follow-up after first treatment
  only Phase 2a

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Dongguk University Medical Center, Ilsan
  - Seoul National Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided